CLINICAL TRIAL: NCT07338851
Title: Evaluation on the Persistence of Sabin Strain Inactivated Poliovirus Vaccine (Vero Cell), Combined Live Attenuated Measles, Mumps and Rubella Vaccine and Freeze-dried Live Attenuated Hepatitis A Vaccine in Chinese Children: Up to 5 Years of Follow-up
Brief Title: the Five-year Antibody Persistence After Immunization With IPV, MMR and HepA-L Vaccines
Status: Not yet recruiting | Type: Observational
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Shaanxi Provincial Center for Disease Control and Prevention (Other); Hubei Provincial Center for Disease Control and Prevention (Other); Jiangsu Provincial Center for Disease Control and Prevention (Unknown); Anhui Provincial Center for Disease Control and Prevention (Unknown); Sichuan Provincial Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Other Study IDs: sIPV/MMR/HepA-L-2025-01
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Polio; Measles; Rubella; Mumps; Hepatitis A
MeSH Terms: conditions — Poliomyelitis; Measles; Rubella; Mumps; Hepatitis A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 5 years of follow-up group: All the children who met the protocol criteria and had been five years since their last doses of sIPV, MMR or HepA-L were included.

SUMMARY:
This study evaluated the antibody persistence of Chinese children five years after they received four doses of sIPV, two doses of MMR vaccine and one dose of HepA-L vaccine.

DETAILED DESCRIPTION:
This is a follow-up study of several previous clinical trials (A Randomized, Controlled, Multicenter Phase 4 Clinic Trial to Evaluate the Immunogenicity and Safety of Combined Immunization of Sabin-strain Inactivated Polio Vaccine (sIPV), Diphtheria, Tetanus, Pertussis Vaccine (DTaP) and Measles, Moms and Rubella Vaccine (MMR) : NCT04054882, NCT04638985; A Randomized, Controlled, Multicenter Phase 4 Clinic Trial to Evaluate the Safety and Immunogenicity of Combined Immunization of Sabin-strain Inactivated Polio Vaccine (sIPV), Diphtheria, Tetanus, Pertussis (DTaP) Vaccine and Live Attenuated Hepatitis A Vaccine (HepA): NCT04053010, NCT04636827). Five years after vaccination with sIPV, MMR or HepA-L, blood samples were collected from the followed-up children to assess the antibody levels and seropositive rates against polio, measles, rubella, mumps and hepatitis A. This study was conducted in six provinces of China.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the NCT04638985 or NCT04636827, and who have completed the vaccination of designated batch numbers of sIPV, MMR or HepA-L vaccines;
* The time window from the day of enrollment to the date when the participants received the fourth dose of sIPV vaccine, the second dose of MMR vaccine, or the first dose of HepA-L vaccine was 60 to 66 months.
* The informed consent form shall be signed by the participant or his/her legal guardian and dated.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have taken part in the NCT04638985 or NCT04636827 trials and have completed the designated batches of sIPV, MMR or HepA-L vaccinations, with a time interval of 60 to 66 months since the fourth dose of sIPV, the second dose of MMR or the first dose of HepA-L vaccination at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
seropositive rates of antibodies against poliovirus | 5 years after the four doses of sIPV immunization
  The percentage of participants with positive antibody(titre ≥ 8) against all three serotypes of poliovirus 5 years after the four doses of sIPV immunization.
seropositive rates of antibodies against measles, rubella, mumps | 5 years after the two doses of MMR immunization
  The percentage of participants with positive antibody against measles, rubella, mumps 5 years after the two doses of MMR immunization.
seropositive rates of antibodies against hepatitis A | 5 years after the one doses of HepA-L immunization
  The percentage of participants with positive antibody against hepatitis A 5 years after the one doses of HepA-L immunization.

SECONDARY OUTCOMES:
GMTs of antibodies against poliovirus | 5 years after the four doses of sIPV immunization
  The GMTs of participants against all three serotypes of poliovirus 5 years after the four doses of sIPV immunization.
GMCs of antibodies against measles, rubella, mumps | 5 years after the two doses of MMR immunization
  The GMCs of participants against measles, rubella, mumps 5 years after the two doses of MMR immunization.
GMCs of antibodies against hepatitis A | 5 years after the one doses of HepA-L immunization
  The GMCs of participants against hepatitis A 5 years after the one doses of HepA-L immunization.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Si County Center for Disease Control and Prevention, Suzhou, Anhui
  - Feixiang District Center for Disease Control and Prevention, Handan, Hebei
  - Sheyang County Center for Disease Control and Prevention, Yancheng, Jiangsu
  - Chenggu County Center for Disease Control and Prevention, Hanzhong, Shaanxi
  - Yanhu District Center for Disease Control and Prevention, Yuncheng, Shanxi
  - Jiangyou Center for Disease Control and Prevention, Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided